CLINICAL TRIAL: NCT03935191
Title: Performance of the Dexcom G6 Continuous Glucose Monitoring (CGM) System in Pregnant Women With Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-903652
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group: Device: Dexcom CGM System
  Interventions: Device: Dexcom CGM System

INTERVENTIONS:
Device: Dexcom CGM System — Dexcom CGM System

SUMMARY:
The purpose of this prospective observational study is to establish the performance and safety of the Dexcom G6 CGM System utilized for up to a 10-day wear period in pregnant women with diabetes mellitus.

DETAILED DESCRIPTION:
Primary Study Objective:

To determine the accuracy of Dexcom G6 CGM System glucose readings in reference to arterialized venous sample YSI glucose measurements in pregnant women with diabetes mellitus.

Secondary Study Objective:

To assess the safety of the Dexcom G6 CGM System, through characterization of device-related Adverse Events (AEs), in pregnant women with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Currently in the 2nd or 3rd trimester of pregnancy;
3. Diagnosis of GDM, T1DM, or T2DM;
4. Willing to avoid insulin injections or wear an insulin pump insertion set within 3 inches from the sensor site;
5. Able to follow study procedures;
6. Able to speak, read, and write in English or Spanish.

Exclusion Criteria:

1. Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
2. Known allergy to medical-grade adhesives;
3. Hematocrit of < 30%;
4. Prescribed tocolytic drugs for treatment of pre-term labor or experiencing high-risk pregnancy complications, including, but not limited to, pre-eclampsia or HELLP syndrome (hemolysis, elevated liver enzymes, and a low platelet count) during current pregnancy;
5. Currently receiving dialysis treatment or planning to receive dialysis during the sensor wear period;
6. Require a Magnetic Resonance Imaging (MRI) scan, Computed Tomography (CT) scan, or diathermy during the sensor wear period;
7. Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study.);
8. Working for a competitive medical device company or having an immediate family member or person living within the same household who works for such a company (e.g., Medtronic, GlySens Inc., Abbott Laboratories, Roche, Senseonics, Waveform, and Ascencia/POCTech);
9. Any condition that, in the opinion of the Investigator, would interfere with their participation in the trial (e.g., marked visual impairment) or pose excessive risk to study staff handling venous blood samples (e.g., known history of HIV or Hepatitis B or C).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age ≥ 18 years;
  2. Currently in the 2nd or 3rd trimester of pregnancy;
  3. Diagnosis of GDM, T1DM, or T2DM;
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Dexcom G6 CGM Accuracy | 10 days
  Accuracy of Dexcom G6 CGM System glucose readings in reference to arterialized venous sample YSI glucose measurements in pregnant women with diabetes mellitus.

SECONDARY OUTCOMES:
Dexcom G6 CGM Safety | 10 days
  Assess the safety of the Dexcom G6 CGM System, through characterization of device-related Adverse Events (AEs), in pregnant women with diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Stayce Beck, Study Director — DexCom, Inc.

IPD SHARING:
Plan to Share IPD: No